CLINICAL TRIAL: NCT06774027
Title: ENCORE: Multicenter ProspectivE Registry of Sequential ANtibody Drug COnjugates (ADCs) in HER2 Negative Metastatic BREast Cancer (MBC)
Brief Title: Prospective Registry of ADC as First- and Second-line Treatment for Breast Cancer
Acronym: ENCORE
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Gilead Sciences (Industry); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 247516; TBCRC 067 (Other: Translational Breast Cancer Research Consortium (TBCRC))
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HER2-negative Breast Cancer; HER2 Negative Breast Carcinoma; Metastatic Breast Cancer; HR+ HER2 Breast Cancer; Metastatic Triple Negative Breast Cancers; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood specimens will be collected during routine clinic visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: HR+/HER2- mBC participants enrolled before first line ADC (ADC1)): Participants with histologically documented HR+/HER2- MBC with a plan to start an FDA-approved ADC as a first ADC per usual care will be enrolled before beginning any ADC. Participants will have blood samples obtained during routine clinical visits during ADC1 and ADC2, if applicable.
  Interventions: Procedure: Specimen collection; Drug: Non-Investigational Antibody-Drug Conjugates (ADC); Other: Medical Record Review
- Cohort 2: Metastatic Triple Negative Breast Cancer (mTNBC) participants enrolled before ADC1: Participants with histologically documented metastatic TNBC with a plan to start an FDA-approved ADC as their first ADC per usual care will be enrolled before beginning any ADC. Participants will have blood samples obtained during routine clinical visits during ADC1 and ADC2, if applicable.
  Interventions: Procedure: Specimen collection; Drug: Non-Investigational Antibody-Drug Conjugates (ADC); Other: Medical Record Review
- Cohort 3: HR+/HER2- mBC Participants enrolled before second line ADC (ADC2)): Participants with histologically documented HR+/HER2- MBC with plan to start an FDA-approved ADC as their second ADC per usual care (ADC1 should be an approved ADC administered per usual care or as monotherapy in a clinical trial; no prior experimental ADCs allowed). Clinical data from the first ADC must be available for retrospective review. Participants will have blood samples obtained during routine clinical visits during treatment of cancer with ADC2.
  Interventions: Procedure: Specimen collection; Drug: Non-Investigational Antibody-Drug Conjugates (ADC); Other: Medical Record Review
- Cohort 4: mTNBC participants enrolled before ADC2: Participants with histologically documented metastatic TNBC with plan to start an FDA-approved ADC as their second ADC per usual care (ADC1 should be an approved ADC administered per usual care or as monotherapy in a clinical trial; no prior experimental ADCs allowed). Clinical data from the first ADC must be available for retrospective review. Participants will have blood samples obtained during routine clinical visits during treatment of cancer with ADC2.
  Interventions: Procedure: Specimen collection; Drug: Non-Investigational Antibody-Drug Conjugates (ADC); Other: Medical Record Review

INTERVENTIONS:
Procedure: Specimen collection — Blood specimens will be collected during regular clinical visits for correlative and exploratory analysis
  Other Names: Biospecimen collection
Drug: Non-Investigational Antibody-Drug Conjugates (ADC) — ADC given under usual care for the treatment of cancer
  Other Names: Non-Investigational ADC
Other: Medical Record Review — Prospective and retrospective medical chart reviews will be conducted to obtain data for analysis.
  Other Names: Medical Chart Review

SUMMARY:
Antibody-drug conjugates (ADCs) have demonstrated substantial improvement in progression free survival (PFS) and overall survival (OS) in phase III clinical trials in patients with metastatic triple negative breast cancer (mTNBC) and hormone receptor positive/HER2 negative (HR+/HER2-) metastatic breast cancer (MBC), offering an effective new treatment strategy. Several outstanding questions drive the decision to use ADC drugs clinically. This is a prospective, multi-site observational study of patients with metastatic breast cancer (mBC) who are being treated with FDA-approved antibody drug conjugates (ADCs) as part of routine care and aims to collect real-world data to evaluate the impact of ADC treatment as part of routine care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Real-world progression free survival (rwPFS) of the first line of ADC under routine care (ADC1) by investigator assessment II. Real-world progression free survival (rwPFS) of the second line ADC under routine care (ADC2) by investigator assessment

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of ADC1 and ADC2 as measured by duration of response (DOR), best overall response (BOR), disease control rate (DCR), and overall survival (OS) for each ADC.

II. To evaluate key safety parameters for ADC1 and ADC2 by chart review.

EXPLORATORY OBJECTIVES:

I. To evaluate/identify correlative biomarkers (e.g., circulating tumor DNA (ctDNA), circulating tumor cells (CTC), and tissue spatial correlates) of response/resistance to ADCs.

II. To evaluate patient reported outcomes (PROs) for each ADC.

OUTLINE:

Participants will have medical chart reviews and biospecimens collected for the duration of routine care with ADC1 and/or ADC2. After the last dose of ADC2, participants will continue to be followed for survival data collection via chart review every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or greater with ability to provide written informed consent for this prospective registry study.
2. Estimated life expectancy of at least at 3 months per investigator assessment.
3. Willingness to provide an archival tissue sample and blood samples (20cc research blood collection at several timepoints) for research purposes.
4. Cohort-specific enrollment criteria:

   * Cohort 1: Histologically documented HR+/HER2- MBC with plan to start an FDA-approved ADC as their first ADC per standard of care (SOC).
   * Cohort 2: Histologically documented metastatic TNBC with plan to start an FDA-approved ADC as their first ADC per standard of care
   * Cohort 3: Histologically documented HR+/HER2- MBC with plan to start an FDA-approved ADC as their second ADC per standard of care (ADC1 should be an approved ADC administered per SOC or as monotherapy in a clinical trial; no prior experimental ADCs allowed). Clinical data from the first ADC must be available for retrospective review.
   * Cohort 4: Histologically documented metastatic TNBC with plan to start an FDA-approved ADC as their second ADC per standard of care (ADC1 should be an approved ADC administered per standard of care or as monotherapy in a clinical trial; no prior experimental ADCs allowed). Clinical data from the first ADC must be available for retrospective review.
   * Measurable disease is not required for any cohort.

Exclusion Criteria:

1. Prior receipt of an experimental ADC in the metastatic setting. Of note, patients who received an FDA-approved ADC as their first ADC (as monotherapy, not in combination) can participate in cohorts 3 or 4 prior to starting their second FDA-approved ADC per standard of care. Of note, for all cohorts, experimental therapies are not allowed as intervening therapies after starting ADC1. If a patient enrolls on a clinical trial of an experimental therapy after ADC1, they will be taken off study.
2. Current participation in a clinical trial with an ADC.
3. Contraindication to research phlebotomy to collect ~20cc blood at each research blood draw timepoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults receiving routine treatment for metastatic breast cancer who have planned, usual care with first line or second line of ADC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-world progression free survival (rwPFS) of first line ADC (ADC1) | Up to 5 years
  rwPFS is defined as the amount of time that elapses between the initiation of ADC1 therapy until the patient experiences disease progression, initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause (whichever comes first).
rwPFS of second line ADC (ADC2) | Up to 5 years
  rwPFS is defined as the amount of time that elapses between the initiation of ADC2 therapy following a previous line of ADC (ADC1) until the participant experiences disease progression, initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause (whichever comes first).

SECONDARY OUTCOMES:
Median Duration of Response (DOR) | Up to 5 years
  DOR is defined as the amount of time between when measurement criteria are met for complete response (CR) or partial response (PR), whichever is first recorded, until the first date that recurrent or progressive disease (PD) is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the usual care ADC began) per Response Evaluation Criteria in Solid Tumors (RECIST) criteria. The participants response will depend on the achievement of both measurement and confirmation criteria.
Best Overall Response (BOR) | Up to 5 years
  The best overall response is the best response recorded from the start of ADC usual care treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The proportion of participants who experience each the following as a best response to usual care ADC: CR, PR, stable disease (SD), PD or not evaluable (NE) per RECIST 1.1 will be reported. The participants best response will depend on the achievement of both measurement and confirmation criteria
Overall Response Rate (ORR) | Up to 5 years
  The ORR is the best response recorded from the start of ADC usual care treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The proportion of participants who experience either CR or PR during usual care ADC will be reported. The participants response will depend on the achievement of both measurement and confirmation criteria
Disease Control Rate (DCR) | Up to 5 years
  The DCR is defined as the proportion of participants who experience complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1 during usual care ADC. The date of first response for either CR, PR, or SD will be used for the calculation of DCR.
Median Real-World Overall Survival Rate (rwOS) | Up to 5 years
  rwOS is defined as the amount of time that elapses between the initiation of usual care ADC and the time of death from any cause, or until the study has completed.
Frequency of usual ADC-related Adverse Events (AEs) | Up to 5 years
  To assess the toxicity profile of each line of usual care ADC, the frequency of key, clinically significant, adverse events by type, grade, ADC line timing, and attribution to each usual care ADC according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Huppert, MD,BA, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be shared with research collaborators